CLINICAL TRIAL: NCT06399614
Title: An Evidenced Based Analytical Study of Occupational Therapy-led Services for Adults Presenting Acutely With a Hand Condition
Brief Title: Occupational Therapy-led Services for Adults Presenting Acutely With a Hand Condition
Status: Recruiting | Type: Observational
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Other Study IDs: ULimerick24
Record Dates: First submitted 2024-03-27; First posted 2024-05-06 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hand Injuries
Keywords: Hand injury; Hand conditions; Occupational Therapy
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention Group: Participants who attend an emergency department or injury unit with access to occupational therapy will be referred to an occupational therapy-led hand therapy clinic. Assessment and intervention for their hand injury will be provided by the occupational therapist, based on existing hand therapy protocols and guidelines. The consultant in charge and the occupational therapist will make clinical judgements with regard suitability for occupational therapy clinics for conservative management of their condition based on patient need at point of triage. Types of interventions provided by the occupational therapist will include customised splinting, targeted exercises and activities, swelling reduction, scar management, desensitisation, education on type of injury, and occupation based intervention. All interventions provided are within occupational therapists' scope of practice and are evidence based.
  Interventions: Other: Occupational Therapy-led Hand Therapy Service
- Care as Usual Group: Participants attending an emergency department of injury unit, do not have access to occupational therapy services and will undergo 'care as usual' in line with the services' protocols and procedures. Care as usual involves standard nursing and medical care and may include: wound care, use of 'off the shelf' orthosis, education, and onward referral to other healthcare professionals.
  Interventions: Other: Care as usual

INTERVENTIONS:
Other: Occupational Therapy-led Hand Therapy Service — Types of interventions provided by the therapist will include splinting, targeted exercises and activities, occupation-based intervention, edema management, scar management; desensitisation, functional tasks completion, and education. All interventions provided are within occupational therapists' scope of practice and are evidence based. Number of treatment sessions will be individualised to the patient and guided by stages of recovery.
  Groups: Intervention Group
Other: Care as usual — Care as usual group: Participants attending an emergency department of injury unit, do not have access to occupational therapy services and will undergo 'care as usual' in line with the services' protocols and procedures. Care as usual involves standard nursing and medical care and may include: wound care, use of 'off the shelf' orthosis, education, and onward referral to other healthcare professionals.
  Groups: Care as Usual Group

SUMMARY:
Traumatic hand injuries account for up to one third of acute hospital presentations. Current guidelines and standards of care recommend patients with hand trauma are seen by hand therapists, typically occupational therapists. The proposed study aims to explore the effectiveness of occupational therapy-led hand therapy services for the adult population presenting acutely to an injury unit or emergency department setting with a hand condition. The research project will consist of an analytical study, involving four different sites in Ireland to enrich findings, and to aid future service development. One site will be the comparison site, as it does not have access to occupational therapy, and will offer patients 'care as usual' upon attendance. Outcome measures will be used for all participants and will be completed at initial patient contact, at week eight and at six months. It is hoped the current proposed study will help shape future service development for those with hand injury including provision of evidence based occupational therapy assessment and intervention.

DETAILED DESCRIPTION:
Traumatic hand injuries account for up to one third of acute hospital presentations. The establishment of Occupational Therapy-led hand therapy clinics is gaining momentum within the literature as improving hand trauma patient care and outcomes. It is identified within the literature that point of acute contact service areas such as accident and emergency or injury unit type settings could benefit from a hand therapy service. The benefits reported include: better patient outcomes, reduced waiting times, reduction of patient presentations to consultant led clinics, faster turnaround of patient care and discharge, reduction of patient complaints, improved patient satisfaction, and reduced costs to the health service.

The proposed study aims to explore the effectiveness of occupational therapy-led hand therapy services for the adult population presenting acutely to an injury unit or emergency department setting with a hand condition. The research project will consist of an analytical study, involving four different sites in Ireland to enrich findings, and to aid future service development. One site will be the comparison site, as it does not have access to occupational therapy, and will offer patients 'care as usual' upon attendance. Outcome measures will be used for all participants and will be completed at initial patient contact, at week eight and at six months. Study objectives include:

1. To define the demographics and characteristics (including functional ability, pain level, and quality of life) of adult service users pre- and post-acute attendance with a hand condition.
2. To profile clinical and process outcomes after initial visit, at 8-week and 6-month follow-up for patients provided with care as usual and those with targeted hand therapy led assessments and interventions.
3. To explore any objective and subjective patient, organizational, and societal benefits of hands service provision.

It is hoped the current proposed study will improve the quality, safety, timeliness and cost of care provided to adults who present to acute services with a hand condition. This information may help shape future service development for those with hand injury including provision of evidence based occupational therapy-led services.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years of age and older
* Adults presenting with an injury and/ or condition of their hand and/or forearm inhibiting function inclusive of: fractures (proximal, middle, and distal phalanx); tendon and soft tissue injury (PIPJ volar plate, central slip +/- lateral band, mallet injury, trigger finger, flexor injury, extensor injury, thumb tendon and ligament injury); digital nerve injury; or carpal tunnel injury.

Exclusion Criteria:

* Patients under 18 years of age
* Patients presenting with complex medical issues in conjunction with a hand injury who may require an alternative pathway, for example, transfer to a different hospital, requiring prioritisation of another medical emergency
* Other exclusions at the discretion of the service depending on team capacity and expertise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years of age and older attending acutely with a hand injury or condition.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Function: our primary outcome is change in patient function for those with acutely presenting hand conditions. | The QuickDASH will be administered at baseline, at 8-weeks (post intervention), and at six months.
  The QuickDASH (Disabilities of the Arm, Shoulder, and Hand) outcome measure is a self report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb. The QuickDASH contains an 11 item disability/symptom scale, with two optional scales capturing sport/art and work ability. The QuickDASH is valid, reliable and has demonstrated high responsive in outpatients with hand trauma and degenerative hand conditions and can be used for clinical and research purposes. A lower score on the QuickDASH denotes lower disability, whilst a high score denotes higher rates of disability.

SECONDARY OUTCOMES:
Change in health related quality of life for those with acutely presenting hand conditions using a visual scale. | The EuroQoL EQ-5D-5L will be administered at baseline, at 8-weeks (post intervention), and at six months.
  The EuroQoL EQ-5D-5L will be used to examine health related quality of life outcomes for patients. This is a standardised measure of health status developed by the EuroQoL group to provide a descriptive profile and an index value for health status. A visual analogue scale reporting respondents self-rated health on a vertical visual analogue scale from 'best imaginable health state' (100) to 'worst imaginable health state' (0) is used to capture self reported change in health related quality of life over time. The visual scale represents the patients perspective and is conceptually different from the index system where a value is attached to a ED-5D-5L profile according to a set of weights that reflect average perspectives on health state.
Change in health related quality of life for those with acutely presenting hand conditions using a descriptive system. | The EuroQoL EQ-5D-5L will be administered at baseline, at 8-weeks (post intervention), and at six months.
  The EuroQoL EQ-5D-5L will be used to examine health related quality of life outcomes for patients. This is a standardised measure of health status developed by the EuroQoL group to provide a descriptive profile and an index value for health status. A descriptive system with five dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression is completed. This part of the outcome tool can be used to generate a health state profile. Each health state can be assigned an index score and analysed against Irish norms. This helps better understand patients health state in relation to each of the five domains as well as being useful for health economic analysis.
Occupational Value and Competence of those with acutely presenting hand conditions. | The Occupational Self Assessment - Short Form (OSA-SF) will be administered at baseline, at 8-weeks (post intervention), and at six months.
  The Occupational Self Assessment - Short Form (OSA-SF) is a validated measure designed to assess one's perceived occupational competence and value, as well as supporting the client by informing goal setting and treatment planning. A higher score denotes higher competence and higher value with performance of occupations, with a maximum score of 48 in the 'competence' subset and 36 in the 'value' subset
Pain reported by those with acutely presenting hand conditions. | The pain verbal rating scale will be administered at baseline, at 8-weeks (post intervention), and at six months.
  A pain verbal rating scale (VRS) will be used to measure pain experience, as rated by the patient with '0' indicating no pain, and '10' indicating worst imaginable pain

CONTACTS AND LOCATIONS:
Overall Officials: Damien Ryan, Principal Investigator — University of Limerick
Locations (5):
- Ireland (5):
  - Beaumont Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - Galway University Hospital, Galway
  - Ennis General Hospital - ULHG, Limerick
  - Nenagh General Hospital ULHG, Tipperary

IPD SHARING:
Plan to Share IPD: No